CLINICAL TRIAL: NCT02283242
Title: Effects of Cholinergic Stimulation on Visceral Fat, Oxidative Stress and Inflammatory Markers in Patients With Metabolic Syndrome: a Randomized Clinical Trial
Brief Title: Galantamine Effects in Patients With Metabolic Syndrome
Acronym: GALANTA-MS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: University of Nove de Julho (Other); Feinstein Institute for Medical Research (Other)
Responsible Party: Principal Investigator, Fernanda Marciano Consolim- Colombo, Fernanda Marciano Consolim Colombo, MD, PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAAE:27386114.9.0000.0068; 2013/22250-9 (Other Grant/Funding Number: Fundação de Amparo à Pesquisa do Estado de São Paulo)
Record Dates: First submitted 2014-10-07; First posted 2014-11-05 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Abdominal Obesity Metabolic Syndrome
Keywords: Cholinergic Antagonists; Inflammation; Oxidative Stress
MeSH Terms: conditions — Abdominal obesity metabolic syndrome; Inflammation | interventions — Galantamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Galantamine (Experimental): * 8 mg of Galantamine for 4 weeks
  * 16 mg Galantamine for 8 weeks
  Interventions: Drug: Galantamine
- Placebo (Placebo Comparator): * 8 mg of placebo for 4 weeks
  * 16 mg placebo for 8 weeks
  Interventions: Drug: Placebo (for galantamine)

INTERVENTIONS:
Drug: Galantamine — Oral use for 12 weeks
  Other Names: Reminyl ER
  Arms: Galantamine
Drug: Placebo (for galantamine) — Oral use for 12 weeks
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
It is recognized that inflammation can be modulated by cholinergic stimulation and that galantamine, an inhibitor of acetylcholinesterase enzyme with central nervous system action, has showed an anti-inflammatory effect, reducing body weight, abdominal fat and improvement in tissue insulin resistance in animal models. Galantamine is a safe drug that is used to treat alzheimer disease.Galantamine treatments of patients with the metabolic syndrome may represent a significant advance in management of this disease. This study aims to investigate the effects of galantamine on inflammatory markers, as well as on abdominal visceral and epicardial fat and oxidative stress in patients with metabolic syndrome. This is a pioneering study that will include expert support. The enrolling of subjects will have continuous monitoring throughout the period of treatment. The study is a double blind randomized prospective study with 60 patients with metabolic syndrome, to be randomized at ratio of 1: 1 placebo and galantamine. The dose of galanthamine is the standard clinically approved (8 and 16 mg). The tracking method include metabolic analysis, inflammatory and oxidative stress markers, hemodynamic evaluation with hear rate variability (sympatho vagal modulation) before, during and after treatment. Computerized tomography assessment of visceral abdominal and epicardial fat before and after treatment will be performed.

DETAILED DESCRIPTION:
Population: patients with metabolic syndrome; Intervention: Galantamine; Comparation: Placebo; Outcomes (primary): proinflammatory cytokines levels.

Description:

Patients with criteria of Metabolic Syndrome (with the 2005 revised NCEP ATP III criteria) will be randomized to 2 groups: use of galantamina (30 patients) or placebo (30 patients) in the following sequency:

I) 4 weeks of treatment with 8 mg of galantamine or placedo (oral ingestion capsules);

II) 8 weeks of treatment with 16 mg of galantamine or placebo (oral ingestion capsules).

Participants will receive a diary to record any symptoms that may present and will be instructed to bring it at each study visit.

Before randomization all participants will go through the following procedures:

* Clinical and neurological evaluation;
* Blood sample analysis of cytokines, oxidative stress and biochemical parameters;
* Multidetector computed tomographic (MDCT) scan of abdomen (visceral - abdominal and epicardial fat) and thorax (calcium score);
* blood pressure recording for hemodynamic evaluation and assessment of heart rate variability
* 24h ambulatory blood pressure measurement

These procedures will be repeated at the end of the protocol.

This is a randomized controlled trial study. Blinding status: Patients, investigators, and outcome assessors.

All participants were outpatients.

The invitation to participate in the study and all the details of the protocol will be explained.

Once the patients have the criteria for inclusion, they receive the cards with capsules containing placebo or galantamine according to continuous numerical order provided by the pharmacy that prepared and randomized such substances (numbered containers).

Drug and placebo will be manipulated and encapsulated in identical packaging at the Central Pharmacy of School of Medicine, University of São Paulo.

We will use simple randomisation using a randomisation table created by computer software - graphpad Software- quickcalcs.

ELIGIBILITY:
Inclusion:

* Diagnosis of Metabolic Syndrome based on recently established criteria (three abnormal findings of the following five)

  * Increased abdominal circumference ≥ 102 cm for men and 90 cm for women
  * Low plasma level of HDL cholesterol < 40md/dL for men and 50 mg/dL for women
  * Increased values for plasma triglycerides > 150 mg/dL
  * Elevated blood pressure ≥130/85 mmHg
  * Elevated level of blood sugar value to 100 mg/dL
* Body Mass Index (BMI) between 25 and 39, with weight maintenance diet and stable for at least 6 months before study entry
* Normal renal function and thyroid function
* Able to participate in the study by signing an informed consent form and comply with study stages throughout its duration

Exclusion:

* On use of antidiabetic medication
* Triglyceride levels ≥ 400 mg/dL or use of lipid lowering medication
* Levels of aspartate transaminase (AST) or alanine transaminase (ALT) ≥ 200 U/L
* Levels of aspartate transaminase (AST) or alanine transaminase (ALT) ≥ 200 U/L
* The office systemic blood pressure ≥160 mmHg or diastolic blood pressure ≥110 mmHg at rest
* BMI ≥ 40kg/m²
* In use of antihypertensive drugs that interfere with the heart rate variability
* On the use of drugs that have known or probable interaction with galantamine: amitriptyline, fluoxetine, fluvoxamine, ketoconazole, oxybutynin, paroxetine, quinidine
* Already participant in regular exercise programs, defined as 90 minutes of activity per week
* Medical history, previous diagnosis or previous supplementary examinations indicating presence of cardiac arrhythmias, coronary artery disease, valvular disease, heart failure, chronic obstructive pulmonary disease, acute or chronic liver disease, renal insufficiency, thyroid disorders, chronic inflammatory diseases, cancer, positive status for HIV, other debilitating diseases
* Abuse of alcohol or other substances in the 12 months prior to study entry
* History of major depression or patients with suicidal ideation
* Personal history of eating disorder
* Utilization of drugs for obesity
* Use of serotonin reuptake inhibitors
* Pregnancy or desire to become pregnant during the study period

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2014-03; Primary Completion 2015-03 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Composite measure of cytokines and adipokines levels, to include IL-1, IL-6, TNF alpha, leptin and adiponectin | 12 weeks

SECONDARY OUTCOMES:
Glucose, triglycerides and high density lipoprotein cholesterol levels | 12 weeks
Insulin levels | 12 weeks
Arterial blood pressure levels | 12 weeks
Heart Rate Variability | 12 weeks
Composite measure of markers of oxidative stress, to include: total amount of free radicals, malondialdehyde, allantoin, anpha-1-antiproteinase, oxidize/reduced glutatione ratio | 12 weeks
Abdominal fat levels | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Fernanda M Consolim Colombo, Dra, Principal Investigator — University of Sao Paulo
Locations (1):
- University of São Paulo, Heart Institute, Medical School, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Consolim-Colombo FM, Sangaleti CT, Costa FO, Morais TL, Lopes HF, Motta JM, Irigoyen MC, Bortoloto LA, Rochitte CE, Harris YT, Satapathy SK, Olofsson PS, Akerman M, Chavan SS, MacKay M, Barnaby DP, Lesser ML, Roth J, Tracey KJ, Pavlov VA. Galantamine alleviates inflammation and insulin resistance in patients with metabolic syndrome in a randomized trial. JCI Insight. 2017 Jul 20;2(14):e93340. doi: 10.1172/jci.insight.93340. eCollection 2017 Jul 20. PMID 28724799